CLINICAL TRIAL: NCT02214186
Title: Impact of Restrictive Fluid Therapy on Renal Function in Severe Preeclamptic Women Submitted to Cesarean Section Under Spinal Anesthesia
Brief Title: Restrictive Fluid Therapy in Severe Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAPPesq 675.011
Record Dates: First submitted 2014-07-16; First posted 2014-08-12 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2014-07

CONDITIONS: Pre-Eclampsia
Keywords: Pre-Eclampsia; Acute Kidney Injury; Fluid Therapy; Anesthesia, Spinal
MeSH Terms: conditions — Pre-Eclampsia; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal Fluid therapy (No Intervention): The liberal group will receive 1500 mL of crystalloid solution during the cesarean section. This is the non-intervention arm once that 1500 ml of crystalloid is the amount usually used during caesarean.
- Restrictive Fluid Therapy (Active Comparator): The restrictive group will receive 250 mL of crystalloid solution during cesarean section.
  Interventions: Other: Restrictive Fluid Therapy

INTERVENTIONS:
Other: Restrictive Fluid Therapy — The intervention in this randomized clinical trial is fluid restriction during cesarean section. The restricted group will receive 250 mL of crystalloid during surgery.
  Arms: Restrictive Fluid Therapy

SUMMARY:
Introduction: Pre-eclampsia is a multifactorial syndrome which occurs in hypertension and proteinuria in pregnant women over 20 weeks gestation. It is the leading cause of maternal complications such as pulmonary edema, which occurs in about 3% of severe preeclamptic having as one of the causes volume overload. Anesthetic procedures are frequent in this population, with replacement with crystalloid of the duct during cesarean section under spinal anesthesia for combat hypotension and hypovolemia manifested by oliguria. However, as water therapy have antagonistic effects on cardiopulmonary and renal systems is no doubt as to the benefits compared to conventional or restrictive pattern of fluid therapy on renal function. Objective: To compare the renal function of patients with severe preeclampsia who received restrictive fluid therapy during caesarean section, as well as evaluating the use of cystatin C and Neutrophil gelatinase-associated lipocalin (NGAL) as a predictor of renal damage in this population. Hypothesis: Intraoperative fluid restriction did not influence renal function of patients with severe preeclampsia undergoing cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
Preeclampsia (PE) is the leading cause of morbidity and mortality worldwide during pregnancy. Fluid therapy for PE women during cesarean section is a controversial issue among medical specialists.

The replacement with crystalloid fluids tool is traditionally used by anesthesiologists during cesarean section under spinal anesthesia for combat hypotension and hypovolemia manifested by oliguria. However, as crystalloid infusion has antagonistic effects on cardiopulmonary and renal systems, there is controversy regarding benefits over conventional and restrictive fluid therapy. Therefore, due to cardiovascular changes in severe PE, restrictive fluid therapy could possibly be beneficial, avoiding complications such as acute pulmonary edema.

Currently, volume replacement during cesarean section in these patients is performed with volumes of about 1500 ml of crystalloid to decrease the chance of developing kidney injury or aggravating previous injury. However, it is not known in the literature whether the renal lesions that appear after birth in patients with PE are just due to the course of the disease itself or can be modified by fluid restriction during the conduct of anesthesia cesarean.

Moreover, intraoperative fluid restriction (250 ml crystalloid) appears as an alternative to handling the patient with PEG, as already safely used in cardiac patients, such as patients with mitral valve stenosis. The security of fluid restriction in patients with PE comes from the fact that pre-eclamptic suffer fewer episodes of hypotension during cesarean section under spinal anesthesia, requiring less fluid input for this purpose. In addition, the pathophysiology of this disease points to a relative hypovolemia, once the delivery performed, with removal of the placenta, fluids kidnapped in excess to third space (tissue edema) will be redirected to the intravascular compartment, restoring homeostasis.

Cystatin C and NGAL (Neutrophil gelatinase-associated lipocalin) arise as valid tools to predict the degree of renal injury. These molecules arise before the onset of renal injury, providing diagnostic and therapeutic actions that can reduce morbidity and mortality related to kidney failure, since some studies have shown that women in first pregnancy with PE are more likely to develop chronic kidney disease that pregnant women without PE.

ELIGIBILITY:
Inclusion Criteria:

* Severe PE was defined as at least one of the following criteria: systolic pressure ≥160 mmHg or diastolic pressure ≥110 mmHg, severe proteinuria (>5 g/24 h), oliguria (<500 ml/24 h), cerebral or visual disturbances, pulmonary edema, epigastric pain, hepatic rupture, impaired liver function, thrombocytopenia, hemolysis, elevated liver enzymes and low platelet count (HELLP) syndrome and evidence of fetal compromise.

Exclusion Criteria:

* previous serum creatinine levels >1 mg/dl
* previous kidney disease
* contraindication to spinal anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wallace A Da Silva, MD, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina da USP; Fernando Bliacheriene, PHD, Study Chair — Hospital das Clínicas da Faculdade de Medicina da USP; Maria José C Carmona, PHD, Study Director — Hospital das Clínicas da Faculdade de Medicina da USP; Carlo Victor A Varela, MD, Study Chair — Hospital das Clínicas da Faculdade de Medicina da USP; Paula C Scherer, MD, Study Chair — Hospital das Clínicas da Faculdade de Medicina da USP; Marcelo Luis A Torres, PHD, Study Director — Hospital das Clínicas da Faculdade de Medicina da USP
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Sibai B, Dekker G, Kupferminc M. Pre-eclampsia. Lancet. 2005 Feb 26-Mar 4;365(9461):785-99. doi: 10.1016/S0140-6736(05)17987-2. PMID 15733721
- [Background] Sibai BM, Mabie WC. Hemodynamics of preeclampsia. Clin Perinatol. 1991 Dec;18(4):727-47. PMID 1764880
- [Background] Aya AGM, Mangin R, Vialles N, Ferrer JM, Robert C, Ripart J, de La Coussaye JE. Patients with severe preeclampsia experience less hypotension during spinal anesthesia for elective cesarean delivery than healthy parturients: a prospective cohort comparison. Anesth Analg. 2003 Sep;97(3):867-872. doi: 10.1213/01.ANE.0000073610.23885.F2. PMID 12933418
- [Background] Pan PH, D'Angelo R. Anesthetic and analgesic management of mitral stenosis during pregnancy. Reg Anesth Pain Med. 2004 Nov-Dec;29(6):610-5. doi: 10.1016/j.rapm.2004.09.006. No abstract available. PMID 15635522
- [Background] Dyer RA, Piercy JL, Reed AR, Lombard CJ, Schoeman LK, James MF. Hemodynamic changes associated with spinal anesthesia for cesarean delivery in severe preeclampsia. Anesthesiology. 2008 May;108(5):802-11. doi: 10.1097/01.anes.0000311153.84687.c7. PMID 18431115
- [Background] Mabie WC, Ratts TE, Sibai BM. The central hemodynamics of severe preeclampsia. Am J Obstet Gynecol. 1989 Dec;161(6 Pt 1):1443-8. doi: 10.1016/0002-9378(89)90901-0. PMID 2603896
- [Background] Dennis AT, Solnordal CB. Acute pulmonary oedema in pregnant women. Anaesthesia. 2012 Jun;67(6):646-59. doi: 10.1111/j.1365-2044.2012.07055.x. Epub 2012 Mar 15. PMID 22420683
- [Background] Aya AG, Vialles N, Ripart J. [Anesthesia and preeclampsia]. Ann Fr Anesth Reanim. 2010 May;29(5):e141-7. doi: 10.1016/j.annfar.2010.03.014. Epub 2010 May 15. French. PMID 20478690
- [Background] Urbschat A, Obermuller N, Haferkamp A. Biomarkers of kidney injury. Biomarkers. 2011 Jul;16 Suppl 1:S22-30. doi: 10.3109/1354750X.2011.587129. PMID 21707441
- [Background] Vikse BE, Irgens LM, Leivestad T, Skjaerven R, Iversen BM. Preeclampsia and the risk of end-stage renal disease. N Engl J Med. 2008 Aug 21;359(8):800-9. doi: 10.1056/NEJMoa0706790. PMID 18716297
- [Background] Xin C, Yulong X, Yu C, Changchun C, Feng Z, Xinwei M. Urine neutrophil gelatinase-associated lipocalin and interleukin-18 predict acute kidney injury after cardiac surgery. Ren Fail. 2008;30(9):904-13. doi: 10.1080/08860220802359089. PMID 18925531
- [Background] Martensson J, Martling CR, Oldner A, Bell M. Impact of sepsis on levels of plasma cystatin C in AKI and non-AKI patients. Nephrol Dial Transplant. 2012 Feb;27(2):576-81. doi: 10.1093/ndt/gfr358. Epub 2011 Sep 12. PMID 21765189
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Derived] Silva WAD, Varela CVA, Pinheiro AM, Scherer PC, Francisco RPV, Torres MLA, Carmona MJC, Bliacheriene F, Andrade LC, Pelosi P, Malbouisson LMS. Restrictive versus Liberal Fluid Therapy for Post-Cesarean Acute Kidney Injury in Severe Preeclampsia: a Pilot Randomized Clinical Trial. Clinics (Sao Paulo). 2020;75:e1797. doi: 10.6061/clinics/2020/e1797. Epub 2020 Jul 22. PMID 32725073

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We calculated the total sample size from a pilot study. Assuming a power of 80% and 95% confidence, the sample necessary to conduct the study was 21 patients in each group of interest. As we considered 10% as maximum margin of loss during follow-up, there were 23 patients enrolled in each group.
Period: Overall Study
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Started | 23 | 23
Completed | 21 | 21
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8) | 33 (5) | 32.07 (6.77)
Gender [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Gestational age (weeks) [Median (Inter-Quartile Range); unit: weeks] | 36.9 [35.3 to 37.0] | 36.7 [30.1 to 37.4] | 36.8 [33 to 37.2]
Body mass index (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 33.78 (7.17) | 31.98 (5.58) | 32.88 (6.37)
Twin pregnancy [Number; unit: participants]
  yes | 2 | 3 | 5
  no | 21 | 20 | 38
Chronic hypertension [Number; unit: participants]
  yes | 11 | 9 | 20
  no | 12 | 14 | 26
Previous preeclampsia [Number; unit: participants]
  yes | 9 | 11 | 20
  no | 14 | 12 | 26
Diabetes Mellitus [Number; unit: participants]
  yes | 9 | 5 | 14
  no | 14 | 18 | 32
Systolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 161 (17) | 170 (20) | 165.5 (18.5)
Diastolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 100.05 (11.75) | 104.80 (15.75) | 102.42 (13.75)

OUTCOME MEASURES:

1. Primary Outcome: Renal Function in Severe Preeclampsia With Restrictive Fluid Therapy
Description: Renal function evaluated through creatinine levels in three moments: preoperative, first and second postoperative days.
Time Frame: preoperative, first and second day postoperative
Population: Were included in the analysis the patients who violated the protocol and lost follow-up (intention to treat analysis)
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Number analyzed (Participants) | 23 | 23
mg/dl
  Creatinine preoperative | 0.69 [0.55 to 0.83] | 0.73 [0.55 to 0.83]
  Creatinine 1st post-operative | 0.99 [0.80 to 1.22] | 0.93 [0.76 to 1.25]
  Creatinine 2nd post-operative | 0.96 [0.80 to 1.09] | 0.84 [0.69 to 1.08]
Statistical Analysis 1: Comparison: Liberal Fluid Therapy vs Restrictive Fluid Therapy; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mann-Whitney followed by Friedman test

2. Secondary Outcome: Neutrophil Gelatinase-associated Lipocalin (NGAL) as New Marker of Renal Injury in Preeclampsia
Description: Evaluate new marker of renal injury (NGAL) in the specific population of patients with severe preeclampsia, comparing the values of first and second postoperative days to baseline.
Time Frame: preoperative, first and second day postoperative
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Number analyzed (Participants) | 23 | 23
mg/L
  NGAL preoperative | 0.16 [0.10 to 0.20] | 0.15 [0.13 to 0.22]
  NGAL 1st post-operative day | 0.18 [0.13 to 026] | 0.21 [0.16 to 0.29]
  NGAL 2nd post-operative day | 0.15 [0.10 to 0.24] | 0.15 [0.11 to 0.22]
Statistical Analysis 1: Comparison: Liberal Fluid Therapy vs Restrictive Fluid Therapy; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mann-Whitney followed by Friedman test

3. Secondary Outcome: Cystatin C as New Marker of Renal Injury in Preeclampsia
Description: Evaluate new marker of renal injury (Cystatin C) in the specific population of patients with severe preeclampsia, comparing the values of first and second postoperative days to baseline.
Time Frame: preoperative, first and second day postoperative
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Number analyzed (Participants) | 23 | 23
mg/L
  Cyst C preoperative | 1.73 (0.6) | 1.99 (0.61)
  Cyst C 1st postoperative day | 1.93 (0.8) | 2.03 (0.66)
  Cyst C 2nd postoperative day | 1.64 (0.5) | 1.72 (0.43)
Statistical Analysis 1: Comparison: Liberal Fluid Therapy vs Restrictive Fluid Therapy; Test type: Superiority or Other; p < 0.05, ANOVA; ANOVA for repeated measures

4. Secondary Outcome: Proteinuria in Severe Pre-eclampsia Submitted to Cesarean Section Under Different Regimes of Hydration
Description: Proteinuria in severe pre-eclampsia submitted to cesarean section under different regimes of hydration. Analyses in pre-operative and post-operative period.
Time Frame: Proteinuria in severe pre-eclampsia in in pre-operative and post-operative period
Measure: Median (Inter-Quartile Range); unit: g/dl
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Number analyzed (Participants) | 23 | 23
g/dl
  Proteinuria pre-operative | 0.46 [0.32 to 1.71] | 2.62 [0.80 to 9.60]
  Proteinuria 1st post-operative day | 0.15 [0.10 to 0.88] | 0.40 [0.28 to 0.58]
  Proteinuria 2nd post-operative day | 0.20 [0.10 to 0.48] | 0.45 [0.10 to 2.23]
Statistical Analysis 1: Comparison: Liberal Fluid Therapy vs Restrictive Fluid Therapy; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mann-Whitney followed by Friedman test

5. Secondary Outcome: Platelets in Restrictive Fluid Management of Severe Preeclampsia
Description: Compare platelets count in the restrictive and liberal groups during the first and second post-operative days.
Time Frame: preoperative, first and second day postoperative
Measure: Mean (Standard Deviation); unit: thrombocytes/mm3
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Number analyzed (Participants) | 23 | 23
thrombocytes/mm3
  Platelets preoperative | 194400 (77867) | 207941 (71371)
  Platelets 1st postoperative day | 183250 (83234) | 201118 (61687)
  Platelets 2nd postoperative day | 192850 (80692) | 221824 (62925)
Statistical Analysis 1: Comparison: Liberal Fluid Therapy vs Restrictive Fluid Therapy; Test type: Superiority or Other; p > 0.05, ANOVA; ANOVA for repeated measures

6. Secondary Outcome: International Normalized Ratio (INR) of Prothrombin Time (PT) in Restrictive Fluid Management of Severe Preeclampsia During Cesarean Section
Description: Compare International Normalized Ratio (INR) of Prothrombin Time (PT) in the restrictive and liberal groups in preoperative, first and second day postoperative.
  PT is expressed in seconds and the entered values represented the INR of PT among study participants and a control population.
Time Frame: preoperative, first and second day postoperative
Population: The values are expressed in seconds and presented as a ration (INR) with control patients.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Number analyzed (Participants) | 23 | 23
ratio
  PT/INR preoperative | 1.00 [0.95 to 1.10] | 0.95 [0.95 to 0.98]
  PT/INR first post-operative day | 1.03 [0.95 to 1.09] | 0.95 [0.95 to 0.99]
  PT/INR seconde post-operative day | 1.0 [0.97 to 1.07] | 0.95 [0.95 to 0.95]
Statistical Analysis 1: Comparison: Liberal Fluid Therapy vs Restrictive Fluid Therapy; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mann-Whitney followed by Friedman test

7. Other Pre Specified Outcome: Urine Output During Cesarean Section in Severe Pre-eclampsia
Description: Urine output during cesarean section in severe pre-eclampsia under two different regimes of hydration (restrictive and liberal)
Time Frame: urine output during cesarean section (an average of 60 minutes)
Measure: Median (Inter-Quartile Range); unit: ml/h
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Number analyzed (Participants) | 23 | 23
ml/h | 116 [69 to 191] | 80 [37 to 110]
Statistical Analysis 1: Comparison: Liberal Fluid Therapy vs Restrictive Fluid Therapy; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Activated Partial Thromboplastin Time in Restrictive Fluid Management of Severe Preeclampsia During Cesarean Section
Description: Compare activated partial thromboplastin time (APPT) and relation with control (R) in the restrictive and liberal groups.
  APPT is a laboratory test that evaluates the efficiency of the intrinsic pathway of coagulation. The unit of measure is seconds and the results are presented as relation (R) with control.
Time Frame: preoperative, first and second day postoperative
Population: The values are expressed in seconds and presented as a ration (R) with control patients.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Number analyzed (Participants) | 23 | 23
ratio
  APPT/R preoperative | 0.98 (0.13) | 1.01 (0.08)
  APPT/R 1st post-operative day | 1.07 (0.10) | 1.03 (0.10)
  APPT/R 2nd post-operative day | 1.07 (0.13) | 1.01 (0.07)
Statistical Analysis 1: Comparison: Liberal Fluid Therapy vs Restrictive Fluid Therapy; Test type: Superiority or Other; p < 0.05, ANOVA; ANOVA for repeated measures

9. Primary Outcome: Postoperative Renal Dysfunction Evaluated by the Acute Kidney Injury Network (AKIN) Index
Description: Renal dysfunction was stratified by the Acute Kidney Injury Network (AKIN) index in three stages, in terms of creatinine increase from baseline: stage 1 included an interval of 150-200%, stage 2 200%-300%, and stage 3 more than 300% or hemodialysis
Time Frame: Postoperative renal dysfunction
Measure: Number; unit: participants
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Number analyzed (Participants) | 23 | 23
participants
  AKIN stage I | 7 | 6
  AKIN stage II | 2 | 4
  AKIN stage III | 1 | 0
Statistical Analysis 1: Comparison: Liberal Fluid Therapy vs Restrictive Fluid Therapy; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Possible adverse event were observed during the first and second post-operative days
Arm/Group | Liberal Fluid Therapy | Restrictive Fluid Therapy
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No